CLINICAL TRIAL: NCT04700280
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered GLPG3970 for 12 Weeks in Adult Subjects With Active Primary Sjögren's Syndrome
Brief Title: A Study Evaluating the Effects of GLPG3970 Given as an Oral Treatment for 12 Weeks in Adults With Active Primary Sjögren's Syndrome (pSS)
Acronym: GLIDER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated based on Sponsor decision
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG3970-CL-207; 2020-003298-22 (EudraCT Number)
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-11

CONDITIONS: Primary Sjögren Syndrome
Keywords: Primary Sjögren Syndrome; Sjögren Syndrome; Autoimmune Diseases; Rheumatic Diseases; Sicca Syndrome
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG3970 (Experimental): Participants will receive GLPG3970 400 milligrams (mg) (2 *200 mg tablet), orally, once daily for 12 weeks.
  Interventions: Drug: GLPG3970
- Placebo (Placebo Comparator): Participants will receive placebo matched to GLPG3970 tablet, orally, once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG3970 — GLPG3970 film-coated tablet.
  Arms: GLPG3970
Drug: Placebo — Placebo film-coated tablet.
  Arms: Placebo

SUMMARY:
This is a first exploration of GLPG3970 in participants with active primary Sjogren's Syndrome (pSS) to evaluate the efficacy, safety and tolerability and to determine its pharmacokinetics (PK) profile compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented diagnosis of pSS for <10 years prior to screening AND defined by the classification criteria >=4 described by the American College of Rheumatology - European League Against Rheumatism (ACR-EULAR).
2. Participant has an ESSDAI score >=5 assessed on 7 domains: constitutional, lymphadenopathy, glandular, articular, cutaneous, hematological, and biological.
3. Participant has an ESSPRI score >=5.
4. Participant has stimulated whole salivary flow rate of >=0.1 milliliter per minute (mL/min).
5. Participant has positive serum titers of anti-Sjögren's-syndrome-related antigen A (anti-SS-A)/Ro and/or anti-SS-B/La antibodies.
6. Participants already on treatment should be on stable standard of care (SoC) for at least 4 weeks prior to first investigational product (IP) dosing.

   The following SoC medications are permitted:
   * Corticosteroids <=7.5 mg/day (prednisone or equivalent); AND/OR
   * Non-steroidal anti-inflammatory drugs (NSAIDs); AND/OR
   * One single antimalarial at a stable dose (hydroxychloroquine <=400 mg/day; quinacrine 100 mg/kg/day, or chloroquine <=250 mg/day); AND/OR
   * One single immunosuppressant at a stable dose (methotrexate [MTX] <=10 mg/week or azathioprine [AZA] <=2 mg/kg/day); AND/OR
   * One single cholinergic stimulant at a stable dose (e.g., pilocarpine, cevimeline).
7. Female participant of childbearing potential must have a negative highly sensitive (serum beta human chorionic gonadotropin or urine dipstick) pregnancy test.
8. Female participant of childbearing potential or male participant must agree to use highly effective contraception/preventive exposure measures.

Key Exclusion Criteria:

1. Secondary Sjögren's syndrome according to the ACR-EULAR (2016) classification.
2. History or presence of unstable condition not related to Sjögren's Syndrome that, in the opinion of the investigator, could constitute an unacceptable risk when taking the IP or interfere with the interpretation of data.
3. Participant has any active systemic infection within 2 weeks prior to first IP dosing, or poorly controlled chronic cardiac, pulmonary, or renal disease.
4. Participant has a known or suspected history of or a current immunosuppressive condition, or a history of opportunistic infections (e.g., human immunodeficiency virus [HIV] infection, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis).
5. Participant has a chronic hepatitis B virus (HBV) infection, as defined by persistent HBV surface antigen (HBsAg) positivity. Participant has hepatitis C virus (HCV) infection, as defined by positive HCV antibody at screening and detectable HCV viremia. Participants with positive HCV antibody must undergo reflex HCV ribonucleic acid (RNA) testing, and participants with HCV RNA positivity will be excluded. Participants with positive HCV antibody and negative HCV RNA are eligible.
6. Participant testing positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as detected at screening based on real time polymerase chain reaction (RT-PCR) or at baseline based on immunoglobulin M (IgM) immunoassay, or participants who have been in contact with SARS-CoV-2 infected individuals in the 2 weeks prior to first dosing of IP. Participants presenting any signs or symptoms of SARS-CoV-2 infection, as detected prior to first IP dosing following careful physical examination (e.g., cough, fever, headaches, fatigue, dyspnea, myalgia, anosmia, dysgeusia, anorexia, sore throat, etc). In addition, any other locally applicable standard diagnostic criteria may also apply to rule out SARS-CoV-2 infection.
7. Participant has taken any disallowed therapies:

   * Mycophenolate mofetil (MMF) within a week prior to screening.
   * Cyclosporine/Tacrolimus within a week prior to screening.
   * Cyclophosphamide within 6 months prior to screening.
   * Ocular medicines (e.g., topical cyclosporine, topical NSAIDs/ corticosteroids) for at least 4 weeks prior to screening, except for a sporadic use.
   * Biologics such as, but not limited to, rituximab, abatacept, and any other unapproved biologic within 6 months prior to screening.
   * Plasmapheresis within 12 weeks prior to screening.
   * Plasma exchange within 12 weeks prior to screening.
   * Intravenous immunoglobulin (IVIG) therapy within 24 weeks prior to screening.
   * Other prohibited medications within 2 weeks or 5 half-lives, whichever is longer, prior to first IP dosing.
8. Concurrent use of anticholinergic agents or any other medication known to cause dry mouth/dry eyes that, in the opinion of the investigator, are a contributing factor to the participant's dryness and/or use of anticholinergic agents not contributing to this dryness, if not stable at least 4 weeks prior to screening.
9. Participant has a history of tuberculosis (TB) diagnosis or evidence of active or latent infection with Mycobacterium tuberculosis.
10. Participant has a history of lymphoma or any malignancy within the past 5 years prior to screening with the exception of excised and curatively treated non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of cervix which is considered cured with minimal risk of recurrence.
11. Participant has severe organ manifestation or life-threatening condition, or has planned a surgery during the study.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Vincent, Study Director — Galapagos NV
Locations (10):
- Universitaetsklinikum Freiburg, Freiburg im Breisgau, Germany
- General Hospital of Athens Laiko, Athens, Greece
- Debreceni Egyetem, Debrecen, Hungary
- Poland (6):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - ETG Lublin, Lublin
  - Centrum Badan Klinicznych S.C., Poznan
  - Medycyna Kliniczna, Warsaw
  - NZOZ Centrum Medyczne Reuma Park, Warsaw
- Medical Center Harmoniya Krasy, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 clinical study sites across 5 countries (1 in Germany, 1 in Greece, 1 in Hungary, 6 in Poland, and 1 in Ukraine).
Pre-assignment Details: A total of 69 participants were screened. Of these, 31 participants were randomized and treated in the study.
Groups:
- GLPG3970: Participants received GLPG3970 400 milligrams (mg) (2 *200 mg tablet), orally, once daily for 12 weeks.
Period: Overall Study
Arm/Group | GLPG3970 | Placebo
Started | 20 | 11
Completed | 9 | 8
Not Completed | 11 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Study terminated by sponsor | 5 | 3
Not completed — Other than specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomized participants who received at least one dose of study drug.
Groups:
- GLPG3970: Participants received GLPG3970 400 mg (2 *200 mg tablet), orally, once daily for 12 weeks.
- Placebo: Participants received placebo matched to GLPG3970 tablet, orally, once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | GLPG3970 | Placebo | Total
Number analyzed (Participants) | 20 | 11 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 10 | 29
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 11 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 11 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ESSDAI Score [Mean (Standard Deviation); unit: score on a scale] — ESSDAI includes 12 domains: constitutional, lymphadenopathy and lymphoma, glandular, articular, cutaneous, pulmonary,renal, muscular, peripheral nervous system, central nervous system [CNS], hematological, biological. Each of the domains was assessed for activity level: no, low, moderate, high. Each domain score was obtained by multiplying the activity level with domain weight (range: 1 to 6), and assigned a numerical score. Sum of all individual weighted domain scores = 0 (best) to123 (worst activity). A higher score indicated more disease activity.
  score on a scale | 12.5 (6.6) | 8.3 (2.4) | 11.0 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in European League Against Rheumatism (EULAR) Sjögren's Syndrome Disease Activity Index (ESSDAI) Score at Week 12
Description: The ESSDAI is a systemic disease activity index to assess 12 domains (organ systems: constitutional, lymphadenopathy and lymphoma, glandular, articular, cutaneous, pulmonary, renal, muscular, peripheral nervous system, CNS, hematological, biological) in participants with pSS. Each of the domains was assessed for activity level (no, low, moderate, and high). Each domain score was obtained by multiplying the activity level with the domain weight, ranged from 1 to 6, and assigned a numerical score based on pre-determined weighting of each individual domain. The sum of all individual weighted domain scores was the overall score, ranged from 0 (best) to 123 (worst activity). A higher score indicated more disease activity. A clinically meaningful reduction from baseline (≥3 points) indicated the improvement of symptoms. Least squares (LS) mean was calculated using mixed models for repeated measures (MMRM).
Time Frame: Baseline, Week 12
Population: Participants in the full analysis set (FAS: all randomized participants who received at least one dose of study drug) with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | GLPG3970 | Placebo
Number analyzed (Participants) | 8 | 5
score on a scale | -4.4 (1.56) | -3.0 (2.03)
Statistical Analysis 1: Comparison: GLPG3970 vs Placebo; Test type: Superiority; p = 0.617, Mixed Models Analysis; LS Mean Difference = -1.4, 90% CI 2-sided [-6.2 to 3.4], Standard Error of Mean 2.69

2. Primary Outcome: Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs) by Severity
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered study drug and which did not necessarily have a causal relationship with study drug. The severity of AEs was graded using the Common Terminology Criteria for Adverse Events (CTCAE) current version at the time of assessment. The maximum intensity of the AE were Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), or Grade 5 (fatal). A TEAE was any AE with an onset date on or after the first dose of GLPG3970 and no later than 30 days after last dose of GLPG3970, or any worsening of any AE on or after the GLPG3970 start date.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (maximum duration=16 weeks)
Population: The safety analysis set included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | GLPG3970 | Placebo
Number analyzed (Participants) | 20 | 11
participants
  Mild | 3 | 4
  Moderate | 5 | 3
  Severe | 3 | 0
  Life-threatening | 0 | 0
  Death | 0 | 0

3. Secondary Outcome: Change From Baseline in EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) Score at Weeks 4, 8, and 12
Description: The ESSPRI is a participant-reported questionnaire to assess subjective participant symptoms and includes 3 domains (dryness, pain, and fatigue). Each domain was scored on scale of 0-10 (0 = no symptom at all and 10 = worst symptom imaginable), and an overall score was calculated as the mean of the 3 individual domains where all domains carry the same weight. Minimum score can be 0 and maximum score can be 10. A higher score indicates worst symptom. A clinically significant reduction from baseline of the ESSPRI score (at least one point or 15% of the baseline value) indicated the improvement of symptoms.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: Participants in the FAS with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | GLPG3970 | Placebo
Number analyzed (Participants) | 19 | 11
score on a scale
  Change at Week 4 | -1.25 (0.37) | -0.60 (0.49)
  Change at Week 8: number analyzed (Participants) | 17 | 8
  Change at Week 8 | -2.05 (0.41) | -1.28 (0.56)
  Change at Week 12: number analyzed (Participants) | 11 | 8
  Change at Week 12 | -2.15 (0.59) | -1.79 (0.70)
Statistical Analysis 1: Comparison: GLPG3970 vs Placebo; Week 4; Test type: Superiority; p = 0.3089, Mixed Models Analysis; LS Mean Difference = -0.64, 90% CI 2-sided [-1.70 to 0.41], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: GLPG3970 vs Placebo; Week 8; Test type: Superiority; p = 0.2834, Mixed Models Analysis; LS Mean Difference = -0.77, 90% CI 2-sided [-1.97 to 0.43], Standard Error of Mean 0.71
Statistical Analysis 3: Comparison: GLPG3970 vs Placebo; Week 12; Test type: Superiority; p = 0.7109, Mixed Models Analysis; LS Mean Difference = -0.36, 90% CI 2-sided [-2.02 to 1.30], Standard Error of Mean 0.95

4. Secondary Outcome: Change From Baseline in ESSDAI Score at Weeks 4, 8, and 12
Description: The ESSDAI is a systemic disease activity index to assess 12 domains (organ systems: constitutional, lymphadenopathy and lymphoma, glandular, articular, cutaneous, pulmonary, renal, muscular, peripheral nervous system, CNS, hematological, biological) in participants with pSS. Each of the domains was assessed for activity level (no, low, moderate, and high). Each domain score was obtained by multiplying the activity level with the domain weight, ranged from 1 to 6, and assigned a numerical score based on pre-determined weighting of each individual domain. The sum of all individual weighted domain scores was the overall score, ranged from 0 (best) to 123 (worst activity). A higher score indicated more disease activity. A clinically meaningful reduction from baseline (≥3 points) indicated the improvement of symptoms. Results of Week 12 is presented in primary outcome measure 1.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: Participants in the FAS with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | GLPG3970 | Placebo
Number analyzed (Participants) | 15 | 7
score on a scale
  Change at Week 4: number analyzed (Participants) | 9 | 6
  Change at Week 4 | -1.7 (1.17) | -1.4 (1.32)
  Change at Week 8 | -3.5 (1.28) | -4.0 (2.02)
Statistical Analysis 1: Comparison: GLPG3970 vs Placebo; Week 4; Test type: Superiority; p = 0.859, Mixed Models Analysis; LS Mean Difference = -0.3, 90% CI 2-sided [-3.6 to 2.9], Standard Error of Mean 1.81
Statistical Analysis 2: Comparison: GLPG3970 vs Placebo; Week 8; Test type: Superiority; p = 0.837, Mixed Models Analysis; LS Mean Difference = 0.5, 90% CI 2-sided [-3.8 to 4.8], Standard Error of Mean 2.46

5. Secondary Outcome: Observed Pre-dose Plasma Concentration (Ctrough) of GLPG3970
Description: Plasma concentration of GLPG3970 observed at pre-dose in nanogram per milliliter (ng/mL), obtained directly from the observed concentration versus time data.
Time Frame: Pre-dose (within 30 minutes prior to dosing) on Weeks 1, 4, 8, and 12
Population: Participants in the pharmacokinetic (PK) analysis set (all randomized participant who received at least 1 dose of study drug and for which plasma concentration data were available) with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GLPG3970
Number analyzed (Participants) | 20
ng/mL
  Week 1: number analyzed (Participants) | 16
  Week 1 | 77.6 (64.7)
  Week 4: number analyzed (Participants) | 15
  Week 4 | 70.4 (108)
  Week 8: number analyzed (Participants) | 9
  Week 8 | 65 (265)
  Week 12: number analyzed (Participants) | 7
  Week 12 | 66 (219)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (maximum duration=16 weeks)
Description: The safety analysis set included all randomized participants who received at least one dose of study drug.
Arm/Group | GLPG3970 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/11
Other Adverse Events (participants affected / at risk) | 10/20 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG3970 (N=20) | Placebo (N=11)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0
Liver injury (Hepatobiliary disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG3970 (N=20) | Placebo (N=11)
Fungal pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Epstein-Barr virus antibody positive (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oral mucosa erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
There were limitations in the dataset, given the small number of participants completing the treatment period due to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators (PI) are NOT employed by organization sponsoring study. There IS an agreement between the PI and Sponsor (or its agents) that restricts PI's rights to discuss/publish trial results after trial is completed. Sponsor must review, approve any results of study or abstracts for professional meetings prepared by investigator(s). Published data must not compromise the objectives of study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT04700280/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT04700280/SAP_001.pdf